CLINICAL TRIAL: NCT01165034
Title: Development,Effectiveness and Cost-effectiveness of a New Respiratory and Palliative Care Out-patient Breathlessness Support Service
Brief Title: Development of King's College Hospital Breathlessness Service
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Irene J Higginson, Professor, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10/H0808/17
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Breathless Patients With Any Established Underlying Medical Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Best usual practice including general respiratory specialist and primary care
- Breathlessness Support Service (Experimental): Patients randomised to the intervention group (IG) will be entered into the BSS in addition to standard best usual care. Expertise in the BSS will comprise of a palliative care consultant or specialist registrar (SpR), a respiratory medicine consultant or SpR with a specialist interest in breathlessness, a respiratory physiotherapist, an occupational therapist and a respiratory nurse specialist. Patients will see 12 health professionals per visit, and multidisciplinary team meetings will take place before and after each visit. Outpatient clinics will take place once per week. The timing of interventions and data collection has been designed to allow for short disease trajectories in patients with cancer and minimise patient burden, whilst allowing time for interventions to have the desired effect. Four weeks is considered to be the minimum length of pulmonary rehabilitation programmes that give a clinically significant benefit.
  Interventions: Other: Breathlessness Support Service

INTERVENTIONS:
Other: Breathlessness Support Service — Patients randomised to the intervention group (IG) will be entered into the BSS in addition to standard best usual care. Expertise in the BSS will comprise of a palliative care consultant or specialist registrar (SpR), a respiratory medicine consultant or SpR with a specialist interest in breathlessness, a respiratory physiotherapist, an occupational therapist and a respiratory nurse specialist. Patients will see 12 health professionals per visit, and multidisciplinary team meetings will take place before and after each visit. Outpatient clinics will take place once per week. The timing of interventions and data collection has been designed to allow for short disease trajectories in patients with cancer and minimise patient burden, whilst allowing time for interventions to have the desired effect. Four weeks is considered to be the minimum length of pulmonary rehabilitation programmes that give a clinically significant benefit.
  Arms: Breathlessness Support Service

SUMMARY:
Breathlessness is a common, distressing symptom in advanced malignant and non malignant disease, and impacts significantly on quality of life. Breathlessness in end stage disease is also responsible for significant healthcare resource usage. Escalante [1] reported hospital admission rates of 60% in patients presenting to a cancer treatment centre with breathlessness. Preliminary trials of breathlessness clinics with selected groups of patients have been promising, but lack data on their cost effectiveness.

The principal aim of the research is to develop and evaluate the effectiveness and cost effectiveness of a multidisciplinary outpatient breathlessness support service (BSS) for the palliation of breathlessness, in advanced malignant and non malignant disease. This is a phase II study that aims to test the hypothesis that a BSS will improve patient mastery over breathlessness and reduce the use of healthcare resources (including GP consultations,accident and emergency attendances, and length of hospital stay) compared with usual best medical care alone (UC),at an acceptable level of cost effectiveness.The outcomes of this study will also help to determine sample size,develop and test methods for a phase III trial that will follow on from this project.

This study will run over 2 years. Breathless patients with advanced malignant and non malignant disease who have already been optimally medically managed will be eligible.

The service will be run in the outpatient department of King's College Hospital, and patients will also be assessed in their own home and by telephone interviews. At baseline we will assess respiratory function and breathlessness mastery and severity using validated scales, and health service usage. Individuals will be randomised to the intervention group [IG] (n=55) or UC (n=55). The IG will attend the new outpatient clinical service with multiprofessional input. Assessments will be repeated at 4, 10 & 24 weeks.

1.Escalante, C.P., Martin, C.G., Elting, L.S. et al., Dyspnea in cancer patients. Etiology, resource utilization, and survival implications in a managed care world. Cancer, 1996. 78(6): p. 13149.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any established underlying medical diagnosis with breathlessness on exertion or at rest.
* Cancer patients who have risk factors for breathlessness( risk factors include a history of smoking, asthma or COPD, lung irradiation, exposure to asbestos, coal dust, cotton dust or grain dust, lung involvement by cancer)
* Respiratory muscle weakness
* Anxiety.
* Patients must have advanced disease that is refractory to maximal optimised medical management. - Patients must be able to engage with a short term physiotherapy and occupational therapy intervention.

Exclusion Criteria:

* Patients with breathlessness of unknown cause.
* Chronic hyperventilation syndrome.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Chronic Respiratory Disease Questionnaire (CRQ) | 12 weeks
  The primary outcome measure will be improvement of mastery of breathlessness, as assessed by a change in the score within the Mastery domain of the chronic respiratory disease questionnaire (CRQ).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Score | Baseline, 6 and 12 weeks during / after the intervention or usual care
A Numerical Rating Scale (NRS) to assess the intensity of the sensation of breathlessness on average and at worst at rest and on exertion over the last 24 hours. | Baseline and 12 weeks post intervention or usual care
Symptom related quality of life(QOL) will also be assessed using the Palliative Care Outcome Scale (POS) and POS symptoms to quantify palliative care symptoms in addition to breathlessness. | Baseline, 6 and 12 weeks during / after the intervention or usual care
EQ5D will be used as a generic health related QOL measure. | Baseline, 6 and 12 weeks during / after the intervention or usual care
  EQ5D is a standardised instrument for use as a measure of health outcome and is especially suited to cost effectivenessanalyses as it can be used to generate qualityad justed life years (QALYs). It is applicable to a wide range of health conditions and treatments, and provides a simple descriptive profile and a single index value for health status.
A subset of patients (10 patients in each treatment group) will undergo qualitative interviews on expectations, and fears about the service. | Baseline, 6 and 12 weeks during / post intervention or usual care
Carer burden will be assessed using the Zarit Burden Inventory. | Baseline, 6, and 12 weeks during / post intervention or usual care
The Client Service Receipt Inventory (CSRI) will be used to record other service use in the three month period prior to baseline assessment and then for each followup period | Baseline, 6 and 12 weeks during / post intervention or usual care
  The CSRI has been used in over 200 studies to assess costs and takes approximately 20 minutes to complete. Services included will be health care (primary and secondary),medication, social care and informal care from family/friends. Lost work time for patients and carers will be recorded.
Physiological status will include forced expiratory volume in 1s, slow vital capacity, peak expiratory flow rate (PEF), and pulse oximetry | Baseline, 6 and 12 weeks durning / post intervention or usual care
Respiratory muscle activity will also be measured noninvasively by quantifying the surface parasternal intercostal muscle electromyogram, to provide an index of neural respiratory drive (NRD). | Baseline, 6 and 12 weeks durning / post intervention or usual care
  This measure is included because disease severity measured by spirometry alone correlates poorly with breathlessness and functional status in respiratory disease. Assessment of NRD using respiratory muscle electromyography provides a measure of the load on the respiratory system, and inclusion of this parameter will provide insights this test in the future phase III trial.

CONTACTS AND LOCATIONS:
Overall Officials: John Moxham, MD FRCP, Study Director — King's College London; Irene Higginson, BMedSci BMBS PhD FFPHM FRCP, Principal Investigator — King's College London
Locations (1):
- King's College Hospital, London, London, United Kingdom

REFERENCES:
- [Derived] Higginson IJ, Bausewein C, Reilly CC, Gao W, Gysels M, Dzingina M, McCrone P, Booth S, Jolley CJ, Moxham J. An integrated palliative and respiratory care service for patients with advanced disease and refractory breathlessness: a randomised controlled trial. Lancet Respir Med. 2014 Dec;2(12):979-87. doi: 10.1016/S2213-2600(14)70226-7. Epub 2014 Oct 29. PMID 25465642
- [Derived] Bausewein C, Jolley C, Reilly C, Lobo P, Kelly J, Bellas H, Madan P, Panell C, Brink E, De Biase C, Gao W, Murphy C, McCrone P, Moxham J, Higginson IJ. Development, effectiveness and cost-effectiveness of a new out-patient Breathlessness Support Service: study protocol of a phase III fast-track randomised controlled trial. BMC Pulm Med. 2012 Sep 19;12:58. doi: 10.1186/1471-2466-12-58. PMID 22992240